CLINICAL TRIAL: NCT01118637
Title: Stepped Care in the Treatment of Trichotillomania
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: American University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, David A. F. Haaga, Professor of Psychology, American University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R15MH086852-01A1 (NIH)
Record Dates: First submitted 2010-05-05; First posted 2010-05-07 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Trichotillomania
Keywords: trichotillomania; self-help; web-based; habit reversal; behavior therapy
MeSH Terms: conditions — Trichotillomania

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate (Experimental): Assigned immediately after baseline assessment to receive step 1 treatment (web-based self-help)
  Interventions: Behavioral: StopPulling.com
- Wait list (No Intervention): Assigned to wait list for 10 weeks before receiving step 1 treatment.

INTERVENTIONS:
Behavioral: StopPulling.com — subsidized access to an interactive self-help website for TTM
  Arms: Immediate

SUMMARY:
Trichotillomania (TTM), repetitive pulling out of one's own hair to the extent that noticeable hair loss occurs, is a distressing condition interfering substantially with functioning and quality of life. The longterm objective of this research is to determine whether psychological treatment of TTM could be disseminated more effectively by using a stepped care model in which less intensive interventions are tried first, with more intensive interventions used only if initial treatment proves insufficient. This project is a pilot study of the first two steps in a stepped care model of treatment. After baseline assessment, 50 participants with TTM will be randomly assigned to (a) Immediate condition, in which they are offered 10-week self-help treatment via an interactive website (Step 1) or (b) Wait List/Delayed Start condition, a 10-week wait list prior to being offered Step 1. In each condition, at the end of Step 1, participants will be offered 8 weeks of in-person habit reversal training provided by psychology graduate students (Step 2). TTM symptoms will be measured from baseline through a follow-up 3 months after the end of Step 2, as will depression, anxiety, quality of life, functional impairment , treatment utilization, and treatment satisfaction.

The specific aims of the study are:

1. To gather preliminary data on the efficacy of web-based self-help, compared to wait list control;
2. To characterize the acceptability of stepped care to patients with TTM by assessing the proportion of enrolled participants who proceed from step 1 to step 2 treatment;
3. To evaluate the convergent validity of four decision rules for concluding that a patient with TTM has benefited sufficiently from a treatment step: (a) No longer meeting TTM diagnostic criteria; (b) Showing a 25% or greater reduction in total scores on self-report and clinician-rated TTM symptoms; (c) achieving complete abstinence from hair-pulling; and (d) clinically significant response on both self-report and clinician-rated TTM symptom measures
4. To evaluate the concurrent and predictive validity of criteria for sufficient benefit from a treatment step by relating them to treatment satisfaction, treatment utilization, and scores on a measure of functional impairment from TTM.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* regular internet access
* if taking medications for Trichotillomania, on stable dose for at least 4 weeks
* have trichotillomania (DSM IV criteria except that increasing and decreasing tension with pulling not required)

Exclusion Criteria:

* current suicidality
* current major depression
* current psychosis
* current severe anxiety
* current substance abuse
* current psychotherapy focused on trichotillomania

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
MGH-HS | 10 weeks
  self-report measure of trichotillomania symptom severity

SECONDARY OUTCOMES:
PITS | 10 weeks
  interviewer rating of trichotillomania symptom severity
Step 2 completion | 18 weeks
  % of patients completing step 1 (self-help) who go on to complete step 2

CONTACTS AND LOCATIONS:
Locations (1):
- American University, Washington D.C., District of Columbia, United States